CLINICAL TRIAL: NCT01621841
Title: Analysis of Visual Pathways in Glaucoma Patients Using a 3tesla-MRI
Acronym: ENVOL
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Union National des Aveugles et DEficients Visuels (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHUBX2012/01
Record Dates: First submitted 2012-06-11; First posted 2012-06-18 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Glaucoma; Fractional Anisotropy
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Glaucoma subjects
- heathly subjects

SUMMARY:
Glaucoma is a neurodegenerative disease representing the second cause of blindness worldwide. IOP (Intra occular pressure) is the most common risk factor, but not the only one as it is observed for normal tension glaucoma. Some studies have reported lesions of the optical pathways on MRI examination MRI 3T (Magnetic Resonance Imaging 3 Telsa), by increasing spatial resolution and DTI (diffusion tensor Imaging)with fractional anisotropy could help us to analyze visual pathways and to determine the association with neurodegenerative diseases as Alzheimer.

The investigators propose to compare volume and structure of the visual pathways between glaucoma patients and healthy subjects matched on age and sex.

Glaucoma is a neurodegenerative disease characterized by loss of retinal ganglion cells, visual field deterioration and optic nerve cupping. Some studies have suggested that all the visual pathways could be damaged in glaucoma. Recently, a German study proved a significant reduction of volume of the optic radiations in glaucoma versus healthy subjects in MRI 3T. Some authors have also suggested that glaucoma could share similarities with the other neurodegenerative diseases like Alzheimer's disease. MRI 3T and DTI allow studying visual pathways with a high level of spatial resolution.Fractional anisotropy is a tag of microstructure.

ELIGIBILITY:
Inclusion Criteria:

* for cases : Age over 40 years-old, glaucomatous lesion of the optic nerve head with cup/disc ratio, visual field loss, and minimental state superior or equal to 28/30
* for healthy subjects/ matched on age and sex, no individual or familial history of glaucoma, IOP less than 21mmHG, minimental state superior or equal to 28/30

Exclusion Criteria:

* Ocular hypertension, optic nerve disease, visual field loss, diabetes, Horton disease, ocular diseases, immunologic diseases, neuropsychiatric diseases, MRI contraindication (pace maker)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Glaucoma subjects are recruted in ophtalmologic departement
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
fractional anisotropy | Inclusion

SECONDARY OUTCOMES:
volume of retrochiasmatic grey matter | Inclusion
global atrophy | inclusion
hyper intensities white matter | inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ophtalmologie Hôpital Pellegrin, CHU de Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Tellouck L, Durieux M, Coupe P, Cougnard-Gregoire A, Tellouck J, Tourdias T, Munsch F, Garrigues A, Helmer C, Malet F, Dartigues JF, Dousset V, Delcourt C, Schweitzer C. Optic Radiations Microstructural Changes in Glaucoma and Association With Severity: A Study Using 3Tesla-Magnetic Resonance Diffusion Tensor Imaging. Invest Ophthalmol Vis Sci. 2016 Dec 1;57(15):6539-6547. doi: 10.1167/iovs.16-19838. PMID 27918827